CLINICAL TRIAL: NCT04662606
Title: Neurofunctional Correlates of Intentional Actions Towards Food Stimuli
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CONSUME
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Food Preferences
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting-group (No Intervention)
- Fed-group (Experimental)
  Interventions: Behavioral: Consumption of a standard meal prior to the fMRI data collection

INTERVENTIONS:
Behavioral: Consumption of a standard meal prior to the fMRI data collection — Consumption of a standard meal prior to the fMRI data collection
  Arms: Fed-group

SUMMARY:
In this project, the investigators will explore the cognitive neuroscience of intentional action in relation to food behaviour. To unravel how the brain systems involved in intentional control of actions and how these interact with the reward system in different physiological conditions and in relation to lean-weight or obesity, the investigators will manipulate the degree of intentionality of the behaviours under examination and the level of satiety of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Normal weight (normal BMI)
* No MRI controindications
* No neurological or cognitive problems

Exclusion Criteria:

* Underweight or overweight
* MRI controindications
* Neurological or cognitive problems

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-09-12 (Actual); Primary Completion 2021-09-12 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
BOLD (Blood Oxygen Level Dependent) signal | This outcome will be measured on the recruitment day
  The investigators will measure the changes of the hemodynamic response (BOLD signal) recorded in the whole brain during the execution of the different experimental tasks (e.g. intentionally guided actions towards stimuli of high or low calories food vs externally guided actions towards stimuli of high or low calories food), in the two groups (fasted and satiated subjects).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Galeazzi, Milan, Italia
  - IRCCS Istituto Ortopedico Galeazzi, Milan, Milano

IPD SHARING:
Plan to Share IPD: No